CLINICAL TRIAL: NCT01820091
Title: An Open Label, Multicenter, Dose Finding, Single Arm, Phase 1 Study of Fusilev® (Levoleucovorin) to Prevent or Reduce Mucositis in Patients With Relapsed or Refractory Non-Small Cell Lung Cancer Receiving Folotyn® (Pralatrexate)
Brief Title: Phase 1 Study of Fusilev® to Prevent or Reduce Mucositis in Patients With Non-Small Cell Lung Cancer Receiving Folotyn®
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPI-FUS-12-103
Record Dates: First submitted 2013-03-21; First posted 2013-03-28 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 10-propargyl-10-deazaaminopterin; Levoleucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 - Fusilev - 20 doses (Experimental): 5 mg/m2 QID (6 hours apart) starting on Days 2 and 16 (24 hours after Folotyn dose) for a total of 20 doses in a 28-day cycle
  Days 2 and 16: 4 doses/day
  Days 3 and 17: 4 doses/day
  Days 4 and 18: 2 doses/day
  Folotyn: 190 mg/m2 on Days 1 and 15 in a 28-day cycle
  Interventions: Drug: Folotyn; Drug: Fusilev
- Cohort 2 - Fusilev - 12 doses (Experimental): 5 mg/m2 BID 8 hours apart on Days 2, 3, 4, 16, 17, and 18 for a total of 12 doses in a 28-day cycle.
  Fusilev dose to start 24 hours after Folotyn dose.
  Folotyn: 190 mg/m2 on Days 1 and 15 in a 28-day cycle
  Interventions: Drug: Folotyn; Drug: Fusilev
- Cohort 3 - Fusilev - 8 doses (Experimental): 5 mg/m2 BID 8 hours apart on Days 2, 3, 16, and 17 for a total of 8 doses in a 28-day cycle.
  Fusilev dose to start 24 hours after Folotyn dose.
  Folotyn: 190 mg/m2 on Days 1 and 15 in a 28-day cycle
  Interventions: Drug: Folotyn; Drug: Fusilev
- Cohort 4 - Fusilev - 4 doses (Experimental): 5 mg/m2 BID 8 hours apart on Days 2 and 16 for a total of 4 doses in a 28-day cycle.
  Fusilev dose to start 24 hours after Folotyn dose.
  Folotyn: 190 mg/m2 on Days 1 and 15 in a 28-day cycle
  Interventions: Drug: Folotyn; Drug: Fusilev
- Cohort 5 - Fusilev - 2 doses (Experimental): 5 mg/m2 once on Days 2 and 16 for a total of 2 doses in a 28-day cycle
  Folotyn: 190 mg/m2 on Days 1 and 15 in a 28-day cycle
  Interventions: Drug: Folotyn; Drug: Fusilev

INTERVENTIONS:
Drug: Folotyn — A cycle of Folotyn treatment is 28 days, with treatment on Days 1 and 15 in each cycle.
  Other Names: Pralatrexate
Drug: Fusilev — Fusilev will be administered either four times a day (QID) (6 hours apart, ±10 minutes), twice a day (BID) (8 hours apart, ±10 minutes) or once a day (QD) by IV push (3-5 minutes) at a dose of 5 mg/m2 according to the cohort to which patients are assigned.
  Other Names: Levoleucovorin

SUMMARY:
To determine the optimal dose and schedule of Fusilev to prevent or reduce Folotyn-related Grade 3 or higher oral mucositis in patients with Non-Small Cell Lung Cancer.

DETAILED DESCRIPTION:
This is an open-label, uncontrolled, nonrandomized, multicenter, dose-finding, single-arm, Phase 1 study primarily to determine the optimal dose and schedule of Fusilev to prevent or reduce Folotyn-related Grade 3 or higher oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Relapsed or Refractory Non Small Cell Lung Cancer (NSCLC) after at least one line of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Histologically or cytologically confirmed Stage III B/IV NSCLC
* Adequate hematological, hepatic, and renal function
* Available during the first 8 weeks of the study treatment period to visit the clinic for oral Mucositis assessments on scheduled days

Exclusion Criteria:

* Active concurrent malignancy. If there is a history of prior malignancies other than those exceptions listed above, the patient must be disease-free for at least 5 years
* Congestive heart failure
* Uncontrolled hypertension
* Known human immunodeficiency virus (HIV)-positive diagnosis
* Previous exposure to Pralatrexate
* Pregnant or breast-feeding women
* Major surgery within 14 days of enrollment
* Active uncontrolled infection, underlying medical condition, or other serious illness that would impair the ability of the patient to receive protocol treatment
* Symptomatic central nervous system (CNS) metastases or lesions for which treatment is required. Patients who received prophylactic CNS treatment are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Optimal dose and Schedule of Fusilev to prevent or reduce Oral Mucositis | Up to 8 weeks
  The study period will begin on the first day of Folotyn treatment (Day 1). Folotyn will be administered intravenously (IV) at a dose of 190 mg/m2 on Days 1 and 15 in a 28-day treatment cycle. Twenty-four hours after the Folotyn dose, Fusilev will be administered either four times a day (QID) (6 hours apart, ±10 minutes), twice a day (BID) (8 hours apart, ±10 minutes) or once a day (QD) by IV push (3-5 minutes) at a dose of 5 mg/m2 according to the cohort to which patients are assigned. Within a given cohort, Fusilev will be administered at the same dose and schedule after each Folotyn dose for the duration of the study.

SECONDARY OUTCOMES:
Impact of Fusilev on the number of Folotyn-related dose modifications secondary to oral mucositis | Up to 8 weeks
  Analysis will involve the number, percent and type of Folotyn dose modification as a function of Fusilev dose.
Impact of Fusilev on the frequency of Oral Mucositis | Up to 8 weeks
  Distribution of the number of cases of oral mucositis will be described by cohort and by degree of mucositis.
Impact of Fusilev on use of Analgesics for Oral Mucositis | Up to 8 weeks
  Oral mucositis assessment form will be provided by the sponsor and is to be completed during treatment visits on day 1 & 15, days 4 &18, end of treatment visits. Patients will complete an Oral Mucositis Daily Questionnaire (OMDQ) starting at Day 1 of Cycle 1 and ending at the End of Treatment visit. Oral mucositis assessment will be assessed in the clinic by the investigator, or designee, and graded according to AE severity as established in the NCI CTCAE scale, Version 4.0.
Impact of Fusilev on number of Folotyn doses delivered | Up to 8 weeks
  All treatment-emergent AEs will be managed per the investigator's judgment or the site's clinical standard of care. Folotyn decrease dose modifications will be made based on Hematologic Adverse Events (absolute neutrophil count) and Non- Hematologic Adverse events (CTCAE v.4) excluding nausea/vomiting for dose adjustments